CLINICAL TRIAL: NCT02852668
Title: Biomechanical Gait Indicators of Elderly Women in Response to Strength Training or Power Training
Brief Title: Power Training Versus Strength Training in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, João Pedro Pinho, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PowerElderly
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: elderly; strength training; power training; functional capacity; gait biomechanics
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Power Training Group (Experimental): Physical exercises. Strength training performed quickly
  Interventions: Other: Power Training
- Strength Training Group (Experimental): Physical exercises. Strength training performed in moderate speed
  Interventions: Other: Strength Training
- Control Group (No Intervention): This group maintained the same physical activity level during the intervention period.

INTERVENTIONS:
Other: Power Training — This experimental groups underwent an intervention period of power training
  Arms: Power Training Group
Other: Strength Training — This experimental groups underwent an intervention period of strength training
  Arms: Strength Training Group

SUMMARY:
The inexorable decline in motor skills during aging provides the investigators with an elderly population with various functional limitations. Among these, the ability to walk, being associated with the risk of falling has been studied by several authors. The adoption of strength and power training as an intervention strategy to reduce the negative effects arising from the physiological or pathological process of aging has been widely discussed in these studies. However, the effects of these interventions on biomechanical gait indicators have not been fully debated yet. Therefore, this study aimed to compare the effects of these two training protocols on functional capacities and biomechanical gait parameters of elderly women.

DETAILED DESCRIPTION:
Three female groups, homogenized by age, body mass index and physical activity level, were formed: the control group (GC: n=8, 69±4 years old), the strength training group (GF: n=6, 67±4 years old) and the power training group (GP, n=7, 68±4 years old). No extra activity was induced to GC's routine. Meanwhile, GF and GP underwent 12 weeks of strength and power training, respectively, with three weekly sessions. While GF performed the exercises with moderate speed (70-90% of 1RM), the GP executed them in fast speed (40-60% of 1RM). A kinematic and electromyographic gait evaluation, as well as balance and functional capacity evaluations, were conducted prior and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* sedentary women with no physical mobility limitations

Exclusion Criteria:

* attending less than 75% of the intervention sessions and not attending the final evaluation

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Gait kinematics | through study completion, an average of 6 months
  toe clearance: minimum vertical distance of the forefoot and the ground during swing phase
Timed up and go test | through study completion, an average of 6 months
  time needed to get up from a seated position walk 3 meters and walk back to the chair
Muscle power | through study completion, an average of 6 months
  knee extensors muscle power
electromyography gait analysis | through study completion, an average of 6 months
  Knee extensors and flexors muscles co-contraction during the gait cycle

CONTACTS AND LOCATIONS:
Overall Officials: Alberto C Amadio, PhD, Study Director — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No
Only group data will be available. These are to be published in scientific papers.